CLINICAL TRIAL: NCT01584375
Title: The Risk of Intraventricular Hemorrhage With Flat Midline Versus Right-Tilted Flat Lateral Head Positions in Preterm Infant Less Than 30 Weeks of Gestation: a Multicenter Randomized Control Trial
Brief Title: The Risk of Intraventricular Hemorrhage With Flat Midline Versus Right-Tilted Flat Lateral Head Positions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low patient recruitment
Sponsor: King Abdul Aziz General Hospital (Other Government)
Collaborators: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Dr. Sameer Al-Abdi, Consultant Neonatologist, King Abdul Aziz General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RE11/022; IRBC/084/12 (Other: KING ABDULLAH INTERNATIONAL MEDICAL RESEARCH CENTER)
Record Dates: First submitted 2012-04-21; First posted 2012-04-25 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2013-11

CONDITIONS: Intraventricular Hemorrhage
Keywords: Intraventricular hemorrhage; Preterm infant; Midline head position; Lateral head Position
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flat midline head position (Other)
  Interventions: Other: Flat midline head position
- Right flat lateral head position (Other)
  Interventions: Other: Right flat lateral head position

INTERVENTIONS:
Other: Flat midline head position — Infant's chin will be kept at a 90±5 degree angle to the bed (the chin and nose being in line with the sternum) throughout the first 168 hours of life.
  --------------------------------------------------------------------------------
  Other Names: FM
  Arms: Flat midline head position
Other: Right flat lateral head position — Infant's head will be tilted 85-90 degrees to right side (approximately the entire chin beyond the right nipple line) throughout the first 168 hours of life.
  Other Names: rFL
  Arms: Right flat lateral head position

SUMMARY:
Intraventricular hemorrhage (IVH) in preterm infants is one of many devastating consequences of prematurity that have both acute and long-term sequelae. Turning a preterm infant's head to one side may increase intracranial pressure and occlude major ipsilateral veins in the neck, which could increase cerebral venous pressure and decrease cerebral venous drainage. Keeping preterm infants' heads in a slightly elevated midline position (side or supine) during the first 168 hours(HOL) has been recommended as one of the 10 potentially better practices to reduce the incidence of IVH in preterm infants. To the best of our knowledge, there has been no systematically collected clinical data quantifying the relationship between IVH and head position in preterm infants. However, the midline head position may challenge the well-known right neonatal head position preference. This preference continues until 3-6 months of age, after which preterm neonates keep their heads mainly in midline. The best head position for preterm neonates is still to be determined. Therefore, the investigators are aiming to conduct a large scale multicenter randomized control trial on order to answer the following research question: Does keeping heads of preterm infants less than 30 weeks of gestation in flat midline (FM) throughout the first 168 HOL reduce the risk of IVH compared to right flat lateral (rFL)? We hypothesized that keeping heads of preterm infants less than 30 weeks of gestation in FM throughout the first 168 HOL would reduce the risk of IVH compared to rFL.

DETAILED DESCRIPTION:
Investigators will randomly assign infants lying on flat (zero degree) beds to be cared for either in a supine FM or a supine rFL head position throughout the first 168 HOL. Investigators will mount a sign on the incubator indicating the assigned head position to be maintained during the first 168 HOL. The goal is to keep the neonates' heads in their assigned positions throughout the first 168 HOL unless a medical indication required a change in position. The left flat lateral head position will be the back-up position whenever the medical conditions of the study neonates preclude maintaining the assigned head positions. The bedside nurse will check the correctness of the infants' head positions every 4 hours by using the built-in spirit (bubble) level of the open-bed incubators and an L-shaped ruler. Investigators are going to use an elbow connector of HUDSON RCI circuit (adult circuit) in a case SENSORMEDICS will be required for neonates in FM group. Investigators will watch and record pressure ulcers or technical difficulties arising from using high-frequency ventilation (HFV) in the infants in FM position. After their first 168 HOL, the study infants will be given routine nursing care provided in their NICU, including a change in head position every 6-12 hours or as needed on a slightly elevated bed. For obvious reasons, the medical team will be unmasked to the assigned head position. It will be left for the physician discretion for controversial/diversity issue (s) in neonatal care but it will be recorded.

Timing of HUS examinations

1. All study neonates will have two screening head ultrasounds (HUS) as follows:

   1. Within first 12 HOL.
   2. At about 168 HOL.
2. Otherwise, investigators will carry HUS according to established IVH diagnosis guidelines:

   1. As early as a clinical suspicion of IVH is raised.
   2. When IVH is detected, then a follow up HUS is repeated within 5-7 days later.

Diagnosis of IVH:

Ultrasound technicians or physicians who have been trained to perform HUS will perform a standard set of HUS views through the anterior fontanel with a high-quality modern real-time portable ultrasound machine with appropriate transducers. They will capture at least six coronal and five sagittal planes. Investigators will send a similar digital format copy of these images and earlier images (if any) to the three study pediatric radiologists who will be blinded to the head position assignments. They independently will report the absence or presence, lateralization (right, left or bilateral), extension, and grade of IVH according to Papile's grading criteria. They will send their reports to the principal investigator via email. If their reports are inconsistent, then diagnosis and grading of IVH will be based on the majority or the consensus among them if majority cannot be reached.

Analysis strategy for withdrawal, drop outs, and protocol violations as both of the following when appropriate:

1. Intention to treat analysis.
2. Per protocol analysis: Including only neonates who will have normal first 12 hours of life HUS, complete the study or develop IVH during the study period, and have their heads kept in the assigned head positions throughout study period (first 168 HOL)or until time of IVH diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Born at the three study NICUs.
2. Gestational age < 30 weeks.

Exclusion Criteria:

1. Lethal congenital anomalies.
2. Hypoxic ischemic encephalopathy.
3. Need external cardiac compression or epinephrine administration at birth.
4. Outborns.

Ages: 1 Hour to 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
All grade IVH incidence | First 168 hours of life.
  To compared all grade IVH incidence in a FM head position with that of a rFL head position in preterm infant less than 30 weeks of gestation.

SECONDARY OUTCOMES:
Severity of IVH | First 168 hours of life.
  To compare Severity of IVH in a FM head position with that of a rFL head position.Investigators will calculate severity score of IVH according to our recent proposed (Al-Abdi 2011).* This proposed severity score is equal to the squared IVH grade of the worse side, plus the IVH grade of the other side, plus 5 for each hemisphere when it has extensive parenchymal involvement (> 2 brain territories), and plus 5 when there is a brain midline shift.
  * Al-Abdi SY. A severity score for intraventricular hemorrhage in preterm neonates. Saudi Med J. Dec 2011;32(12):1313-1314.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in:
  1. Preterm infants less than 28 weeks of gestation.
  2. Singletons.
  3. Multiple gestations.
  4. Neonates who will complete the study, have normal first 12 hours of life HUS, and their heads will be kept in the assigned head positions of at least 85% of study duration.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 24-47 hours of life.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 48-71 hours of life.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 72-95 hours of life.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 96-119 hours of life.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 120-143 hours of life.
Subgroup analysis | First 168 hours of life.
  To compare all grade IVH incidence at about 168 HOL in a FM head position with that of a rFL head position in neonates who will have normal first 12 hours of life HUS and their heads will be kept in the assigned head positions for the first 144-167 hours of life.
Complications | First 168 hours of life.
  To compare incidence of: 1) Pressure ulcer as per calcification of the National Pressure Ulcer Advisory Panel (NPUAP) and ; 2) pressure alopecia in a FM head position with that of a rFL head position.
Diagnosis of IVH | First 168 hours of life
  Progression of IVH which will be diagnosed within the first 12 HOL.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Al-Abdi, SSCP, FRCPCH, Principal Investigator — King Abdulaziz Hospital
Locations (3):
- Saudi Arabia (3):
  - Almana General Hospital, Al-Ahsa, Eastern Province
  - King Abdulaziz Hospital, Al-Ahsa, Eastern Province
  - King Abdulaziz Medical City, Jeddah, Mecca Region